CLINICAL TRIAL: NCT02253355
Title: PINS Stimulator System for Patients With Treatment Resistant Depression
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-006
Record Dates: First submitted 2014-09-27; First posted 2014-10-01 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Treatment-Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Experimental): Stimulation is on
  Interventions: Device: Deep Brain Stimulation
- Placebo (Sham Comparator): Stimulation is off
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation
  Other Names: PINS Stimulator System

SUMMARY:
Evaluate the effects and safety of Deep Brain Stimulation (DBS) to treat on patients with Treatment-Resistant Depression (TRD) and using functional magnetic resonance imaging (fMRI)to evaluate the influence of acupuncture on patients, which will be afford objective evidence for the mechanism of Acupuncture on depression.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ages 20-70 years
2. Diagnosed with non-psychotic major depressive disorder, single or recurrent episode by DSM-IV-TR criteria
3. First episode onset before age 45
4. Current episode > 12 months duration
5. In the current episode: Documented resistance (i.e. persistence of the major depressive episode) to a minimum of 4 adequate depression treatments from at least 3 different treatment categories (e.g. SSRI's)
6. SNRI's, TCA's, MAO-inhibitors, Mirtazipine, Nefazodone, Trazodone, Bupropion, lithium augmentation, thyroid augmentation, ECT); Adequacy of treatments as defined by a score of at least 3 according to the amended Antidepressant Treatment History Form (ATHF) criteria
7. Hamilton Depression Rating Scale (HDRS) of > 20 at 3 separate baseline visits, rated by 2 separate psychiatrists, Baseline 2 and Baseline 3 HDRS scores cannot improve ≥ 25%

Exclusion Criteria:

1. Patients with hearing impairment
2. Failures of important organs and in severe conditions
3. Be reluctant or disabled to receive neuropsychological assessments;
4. Participate in other clinical trial
5. Has a life expectancy of < 1 year
6. The investigator and/or enrollment review committee, would preclude participation in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the Hamilton Depression Rating Scale-17 | 1, 3, 6 and 12 months of stimulation

SECONDARY OUTCOMES:
The incidence of all adverse events | 1, 3, 6 and 12 months of stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Li Luming, PhD, Study Chair — Tsinghua University